CLINICAL TRIAL: NCT01170767
Title: French Evaluation Group Avastin Versus Lucentis
Acronym: GEFAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007.467/10
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2013-02

CONDITIONS: Age Related Macular Degeneration
Keywords: Age-related Macular Degeneration; Bevacizumab; Ranibizumab
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Avastin (Experimental): intravitreal injection of bevacizumab
  Interventions: Drug: Avastin
- Lucentis (Active Comparator): intravitreal injection of ranibizumab
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: Avastin — Intravitreal injection of bevacizumab at a concentration of 1.25 mg per injection. One injection per month at the maximum and between 3 and 12 injection in the whole study.
  Arms: Avastin
Drug: Lucentis — Intravitreal injection of ranibizumab at a concentration of 0.50 mg per injection. One injection per month at the maximum and between 3 and 12 injection in the whole study.
  Arms: Lucentis

SUMMARY:
Age Related Macular Degeneration (AMD) is the first cause of visual impairment in elderly patients in industrialized countries. Neovascular or "wet" AMD, characterized by the presence of choroïdal neovessels, represents the most aggressive form of the disease. Its prevalence is 3.3% among patients older than 65 years in Europe, and increases with age.

Intraocular injections of anti-angiogenic monoclonal antibodies (ranibizumab) to treat AMD have appeared recently. It is derived from a larger sized molecule, bevacizumab, which do not have the market authorization for this indication. However, numerous publications of case series seem to show the effectiveness and a satisfactory safety profile of bevacizumab.

These conclusions have to be confirmed with a high level of evidence study. The aim of the GEFAL study is to demonstrate non-inferiority of effectiveness in clinical terms after 12 months of treatment with bevacizumab compared to ranibizumab on the visual acuity of patients affected by neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years old
* Affected by neovascular retrofoveal AMD whatever the subtype, unilateral or bilateral (the eye included will be chosen by the investigator and the patient);
* Best corrected VA for the studied eye ranging between 20/32 (6.3/10) and 20/320 (0.6/10) with ETDRS scale
* Size of lesion < 12 disk area
* In case of occult neovessels, proof required of recent development of the lesion: loss of VA of at least 5 letters ETDRS (equivalent one line) in the last 3 months OR appearance of a subretinal heamorrhage OR increase in the size of the lesion (> 10%) using fluoresceinic angiography during the last month by comparison with the last 3 months OR appearance of OCT criteria of macular oedema type, serous separation of neuro-epithelium, separation of the pigmented epithelial during the last month
* Effective birth control for sexually active female
* Signed informed consent.

Exclusion Criteria:

* Previous or actual treatment with intravitreal injection of an anti-VEGF drug (ranibizumab, bevacizumab or pegaptanib) in the studied eye
* Other healing treatment in the studied eye during the last 3 months before the first injection
* Medical history of photocoagulation in the studied eye
* Involvement in another clinical study (studied eye and/or the other eye)
* Subretinal haemorrhage reaching the fovea centre, with a size > 50% of the lesion area
* Fibrosis or retrofoveal retinal atrophy in the studied eye
* Retinal pigment epithelial tear reaching the macula in the studied eye
* Choroidal neovascularisation not related to a DMLA in the studied eye
* Medical history of intravitreal medical device in the studied eye
* Active or suspected ocular or peri-ocular infection
* Serious active intra-ocular inflammation in the studied eye
* Medical history of auto-immune or idiopathic uveitis
* Proved diabetic retinopathy
* Intra-ocular pressure ≥ 25 mmHg despite two topical hypotonic treatments
* Medical history of intra-ocular surgery within 2 months before the first injection in the studied eye
* Aphakia or lack of lens capsule (not removed by YAG laser) in the studied eye
* Any illness or ocular condition that would require an intra-ocular surgery in the studied eye within 12 months after the inclusion
* Known hypersensitivity to ranibizumab, bevacizumab, or another drug composite of the medicinal products used; allergy to fluorescein, indocyanin green, anaesthetic eye drops
* Arterial hypertension that is not controlled by an appropriate treatment
* Previous or actual treatment with systemic administration of bevacizumab
* Follow up not possible during 12 months
* No affiliation to the French national health insurance program.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the mean change from inclusion to 12 months post initiation of treatment in VA score, measured on the "Early Treatment Diabetic Retinopathy Study" (ETDRS) scale at an initial distance of 4 meters. | 12 months

SECONDARY OUTCOMES:
Evaluate and compare the efficacy of treatments by bevacizumab and ranibizumab | 12 months
Evaluate and compare the proportion of adverse events occurring at the local and systemic level in the two groups. | 12 months
Describe and compare the dosage regimen (average number of injections and time before re-injection) in the two groups | 12 months
Describe the pharmacokinetic profile of the drugs in blood and aqueous humor in a sub-group of 20 patients, during the induction stage. | 3 months
Create a medico-economic model of the impact related to the two strategies. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent KODJIKIAN, Principal Investigator — Hospices Civils de Lyon - Hôpital de la Croix-Rousse
Locations (1):
- Service d'Ophtalmologie - Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Kodjikian L, Souied EH, Mimoun G, Mauget-Faysse M, Behar-Cohen F, Decullier E, Huot L, Aulagner G; GEFAL Study Group. Ranibizumab versus Bevacizumab for Neovascular Age-related Macular Degeneration: Results from the GEFAL Noninferiority Randomized Trial. Ophthalmology. 2013 Nov;120(11):2300-9. doi: 10.1016/j.ophtha.2013.06.020. Epub 2013 Aug 2. PMID 23916488